CLINICAL TRIAL: NCT00261625
Title: Can Alendronate Suppress Aortic and Coronary Artery Calcification and Improve Bone Mineral Density in Chronic Peritoneal Dialysis Patients?
Brief Title: Can Alendronate Suppress Calcification and Improve Bone Density in Chronic Peritoneal Dialysis Patients?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 940706
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: End-Stage Renal Disease; Osteoporosis
Keywords: peritoneal dialysis; artery calcification; bone mineral density
MeSH Terms: conditions — Kidney Failure, Chronic; Osteoporosis | interventions — Alendronate

INTERVENTIONS:
Drug: alendronate

SUMMARY:
Alendronate is a safe and effective drug for treating osteoporosis in post-menopausal women. However, its safety and efficacy in increasing bone mineral density in chronic peritoneal dialysis (PD) patients have not been investigated. Etidronate, another bisphosphonate, can suppress the extent of coronary artery calcification in chronic hemodialysis patients. The hypothesis of this study is that alendronate can increase bone mineral density and suppress aortic and coronary artery calcification in chronic peritoneal dialysis patients.

DETAILED DESCRIPTION:
Study Design

The study is a prospective, randomized cross-over study. Fifty patients will be included. All participants are randomly allocated to either group 1 or group 2. Each group consists of 25 patients. Group 1 patients receive alendronate 70 mg once weekly in the first 24 weeks of the study, while group 2 patients receive the same dose of drug every week in the second 24 weeks. The extent of coronary artery and aortic calcification is evaluated by using multidetector spiral computed tomography, whereas bone mineral density is measured by dual-energy X-ray absorptiometry. Both examinations are performed at week 0, 24 and 48 for each participant. Serum level of calcium should be kept within normal limits and serum level of phosphorus should be kept below 6 mg/dl.

Administration of Alendronate

One tablet of alendronate (70 mg per tablet) should be swallowed by each patient once every week with water at least 30 minutes before breakfast, beverage or medication of the day during the treatment period. Patients must not lie down for at least 30 minutes after taking the drug.

Measurement of Coronary Artery and Aortic Calcification

Multidetector spiral computerized tomography (CT) of the chest is performed at week 0, 24 and 48 for each participant to measure the extent of coronary and aortic calcification.

Measurement of Bone Density

Dual energy X-ray absorptiometry is performed at week 0, 24 and 48 for each participant to measure the density of bone.

Demographic and Clinical Characteristics of Patients

Patients characteristics such as age and sex are documented. Clinical parameters including body height, body weight, duration of dialysis, calcium concentration of dialysate, and medication under use are recorded. Blood pressure is measured at each clinical visit for 3 times after the patient has sit for at least 15 minutes.

Collection of Laboratory Data

Fasting serum levels of albumin, phosphorus, calcium, alkaline phosphatase (ALP), intact parathyroid hormone (iPTH) and hemoglobin level of each patient are checked at study entry and once every month. Fasting serum levels of triglyceride, total cholesterol, high-density lipoprotein cholesterol (HDL-chol), low-density lipoprotein cholesterol (LDL-chol), and hypersensitive C-reactive protein (CRP) of each patient are checked at study entry and once every 3 months.

Record of Adverse Effects of Alendronate

Any adverse effect of alendronate is recorded every month at clinic visit.

Compliance of Patients

Compliance of the patients is monitored using telephone calls once every week during the treatment period with alendronate.

ELIGIBILITY:
Inclusion Criteria:

1. Have received maintenance PD for more than 3 months at National Taiwan University Hospital,
2. Have high CPP level (≧50), and
3. Have chest X-ray proven aortic calcification or coronary artery calcification proven before.

Exclusion Criteria:

Patients are excluded if they have any one of the following conditions:

1. Had been hospitalized in recent 3 months due to severe comorbid diseases,
2. Are hypersensitive to alendronate or any of its components,
3. Have esophageal diseases
4. Are not able to stand or sit upright for 30 minutes,
5. Have refractory hypocalcemia, or
6. Patients who are pregnant.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
extent of aortic and coronary artery calcification with and without the use of alendronate
bone mineral density with and without the use of alendronate

SECONDARY OUTCOMES:
serum levels of calcium, phosphorus and parathyroid hormone

CONTACTS AND LOCATIONS:
Overall Officials: Tze-Wah Kao, Master, Principal Investigator — National Taiwan University

REFERENCES:
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877